CLINICAL TRIAL: NCT04373447
Title: Laparoscopic Cholecystectomy is no More Risky in Emergent Cases With in Cardiopulmonary Risk: Fundus-Callot Cholecystectomy With Low Pressure Pneumo-peritoneum VS Open Cholecystectomy - Randomized Controlled Trials
Brief Title: Laparoscopic Cholecystectomy is no More Risky in Emergent Cases With in Cardiopulmonary Risk: Fundus-Callot Cholecystectomy With Low Pressure Pneumo-peritoneum VS Open Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lap cholecystectomy 2
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fundus-calot laparoscopic cholecystectomy (Active Comparator): use laparoscopic fundus first then calot dissection cholecystectomy
  Interventions: Procedure: lap fundus-calot cholecystectomy
- open cholecystectomy (Active Comparator): open cholecystectomy
  Interventions: Procedure: open cholecystectomy

INTERVENTIONS:
Procedure: lap fundus-calot cholecystectomy — use laparoscopic fundus-calot approach
  Arms: fundus-calot laparoscopic cholecystectomy
Procedure: open cholecystectomy — use open approach
  Arms: open cholecystectomy

SUMMARY:
Introduction:

In the last decades and due to improvement of medical heath care, large number of elderly persons were prevalence. Old age usually had cardiopulmonary different diseases. Biliary problems are high in old age. advancement of laparoscopic that occurred in the last years made the use of laparoscopy is available in these cardiopulmonary risk patients. many studies faced the role of laparoscopy in acute cholecystitis in elderly but no studies stated a new and a safe laparoscopic approach to the patients.

Aim: compare between Fundus-Calot cholecystectomy with low pressure pneumo-peritoneum VS open cholecystectomy in Emergency cases with cardiopulmonary risk patients as regard intraoperative data and postoperative complications.

Patients and methods:

This study prospective randomized controlled study was conducted on 374 cases with acute cholecystitis, biliary colic, mucocele and pyocele of gall bladder in emergency general surgery department. Patients were divided into 2 groups, Group A: fundus-Calot approach (235cases) and Group B (235cases): classical open approach

DETAILED DESCRIPTION:
1. INTRODUCTION Evolving the role of laparoscopy in the last decades in managing of different surgical diseases especially biliary diseases had made laparoscopic cholecystectomy of special interest in the field of surgery. The wide spread of use of laparoscopic cholecystectomy put this surgery in the front line of the commonest operation performed in digestive system surgery and really put open cholecystectomy a side.[ Gouma DJ, Rauws EA, Lameris JS. Bile duct injury after cholecystectomy: risk of mortality substantially higher. NedTijdscr Genseeskd 2004; 148: 1020-24.]

   Laparoscopic cholecystectomy advantages are numerous to both the doctors and the patients. Advantages to the surgeons are safety and rapidity of the operation with experienced surgeons. To the patients as regard small sized operative wounds, less pain postoperative, less wound infection and hence rapid discharge from hospital and regain its usual daily activities . [Stanisic V, Bakic M, Maqgelinic M, Kolasinac H. Babic I. [Laparoscopic cholecystectomy of acute cholecystitis]. Med Preql 2010; 63: 404-8.]

   Despite the fact that laparoscopic approach had many benefits over open approach, yet many hazards may occur from laparoscopic cholecystectomy starting with viscous injury during induction of pneumoperitoneum and conversion till fatal biliary and vascular injuries during blind and insisted dissection of disturbed anatomy and frozen Calot triangle. these complications may occur with best surgical hands and decreased with increasing learning curve.[ Russel JC, WalshSJ, Mattie AS, Lynch JT. Bile duct injuries.1989- 1993: A state wide experience: Connecticut laparoscopic cholecystectomy registry. Arch Surg 1996; 131:382-8.][ Atmaram DC, Lakshman K. Predictive factors for conversion of laparoscopic cholecystectomy. Indian J Surg 2011; 73: 42-3] a study put us on the way to avoid bile duct injuries [5].

   The incidence of gall bladder disease increase with advancement of age so that 20-30% of patients undergo laparoscopic cholecystectomy is elderly patients > 60 years with cardiopulmonary risks. and increase to 80 % after 90 years .Elderly patients had cardiopulmonary risks and reduced physiological reserve [Festi D, Dormi A, Capodicasa S, Staniscia T, Attili AF, Loria P, et al: Incidence of gallstone disease in Italy: results from a multicenter, population-based Italian study (the MICOL project). World J Gastroenterol 2008; 14:5282-5289.] [Ratner J, Lisbona A, Rosenbloom M, Palayew M, Szabolcsi S, Tupaz T: The prevalence of gallstone disease in very old institutionalized persons. JAMA 1991; 265: 902-903.]. Other study stated lower incidence of acute cholecystitis in the elderly group of only 6%[ S. W. Lee, S. S. Yang, C. S. Chang, and H. J. Yeh, "Impact of the Tokyo guidelines on the management of patients with acute calculous cholecystitis," Journal of Gastroenterology and Hepatology, vol. 24, no. 12, pp. 1857-1861, 2009.]

   Insufflation of CO2 induces both hemodynamic and mechanical effects. Compression of the vascular system decrease cardiac output due to increase peripheral resistance. Abdominal distension hinder movement of diaphragm. [ Enciso NJ (2013) Anestesia en la cirugía laparoscópica abdominal. An Fac med 74(1): 63-70.].

   Head up position during laparoscopic cholecystectomy decrease venous return and release catecholamine in the blood causing increase in peripheral vascular resistance and myocardium exerts more efforts to pump the blood against high peripheral resistance.[13][14] [15]

   No randomized studies have compared fundus-Callot laparoscopic cholecystectomy with low pressure pneumoperitoneum with open cholecystectomy in cardiopulmonary risk patients with urgent cholecystectomy.

   The aim of this study was to evaluate and compare the outcome of urgent LC using either fundus-Callot approach or open approach in cardiopulmonary risk patients as regard morbidity and mortality.
2. THE AIM OF THE WORK The aim of this study was to evaluate and compare the outcome of urgent laparoscopic cholecystectomy under low pressure Pneumo-peritoneum using either fundus-Callot first approach Vs open approach in cardiopulmonary risk patients as regard morbidity and mortality.
3. Patients and methods Study design: Prospective Randomized controlled clinical study. Study place: our study was conducted in the surgical emergency unit of our University Hospitals.

Study period: March 2015 to March 2018. Source of data: Patients admitted with clinical diagnosis of acute cholecystitis, biliary colic, mucocele or pyocele of gall bladder in patients with cardiopulmonary diseases.

Sample size: A total of 374 patients with a clinical diagnosis of acute cholecystitis, biliary colic, mucocele or pyocele of gall bladder in patients with cardiopulmonary diseases.

Sampling method: simple random sample with a balance the data were uploaded into the database using a standard closed-field electronic form; to guarantee patient anonymity, no information that could permit patient identification was registered in the database.

Method of sample size calculation: Sample size calculated to be 187 at each group based on global complications rate difference between open and laparoscopic group from previous paper with 80% power of study and 95% confidence interval

Patient selection criteria:

A. Inclusion criteria:

1. Age: any age.
2. Sex: Male and Non pregnant female.
3. Patients with cardiopulmonary diseases.
4. Patients who diagnose acute cholecystitis not improving on medical treatment for 48 hours.
5. Patients with biliary colic, mucocele of gall bladder and pyocele of gall bladder.
6. American Society of Anesthesiologist's (ASA) score: grade I, II, III.

Exclusion criteria:

1. ASA grade IV
2. Patients refuse surgery.
3. Documented neurological, renal and Liver disease.
4. Previous percutaneous cholecystostomy
5. Cases not tolerated CO2 insufflation from the start.
6. Other associated problems as acute cholangitis, pancreatitis, gastro-intestinal cancer or bile duct diseases

Preoperative work up: All patients included in the study underwent:

1. Full clinical examination: pain in right hypochondrium radiated to right shoulder, local examination revealed tenderness in right hypochondrium or mass and fever.
2. Ultrasonography: thick edematous wall of gall bladder distended gall bladder or stone impacted in gall bladder neck.
3. Blood investigations :leukocytosis
4. Liver Function Tests.
5. Chest x-ray and pulmonary function test.
6. ECG and Echocardiography.

The patients are admitted to the ward where third generation cephalosporin, metronidazole, pethidine, proton pump blockers and intravenous fluid were started.

Patients are divided into 2 groups:

Group A (n=187): patients underwent laparoscopic cholecystectomy with low pressure pneumoperitoneum and initial fundus first cholecystectomy followed by dissection of Calot triangle (fundus-Calot dissection) Group B (n=187): patients underwent open cholecystectomy

Efforts to decrease bias in the study:

1. For pretrial bias: Good Define objectives. Risk and outcome .Select patients on probability sample with adequate sample size. Define confound factors and avoid it
2. To avoid during trial bias: Standardize reaction and management of patients blindly-Objective data use rather than subjective-Good handling of data- plan designed for drop out
3. To avoid after trial bias: Suitable statistical analysis used-Good and carefully interpretation-Control of confound

Methods:

The patients were given general anesthesia. The stomach and the urinary bladder were deflated with naso-gastric tube and a catheter. The anaesthiologist continuously monitor the vital signs, PO2 and PCO2 of the patients throughout the surgery. Insufflation of the abdomen were done by either Verres needle or open Hasson techniques. Endoscope was introduced through the umbilical incision and the other three trocars were introduced in epigastrium(10 mm), right subcostal(5 mm) and right anterior axillary line at the level of umbilicus(5mm).we started release of the fundus first by incision of the peritoneum on left side of middle of gall bladder, and the dissection continued in the peritoneum around the fundus to the other side in inverted u-shaped figure. Then the fundus of gall bladder is freed from the liver by coagulation. Then the fundus is grasped to the right shoulder with ease and this help elevation of the neck of gall bladder into view. We then begin to dissect the cystic duct and cystic artery with blunt and sharp dissection till critical view of safety appears. The cystic duct and artery are controlled by clips and divided. Finally the rest of gall bladder adherent to the liver is removed. A drain is put in gall bladder bed.

Open cholecystectomy: subcostal Kocher incision. The abdominal layer is entered till opening the peritoneum. By the use of retractors, the neck of gall bladder is exposed and any adhesion from omentum, colon or duodenum is released carefully. Then we dissect on cystic duct and artery carefully and they were controlled by Vicryl 2/0 sutures. Then the gall bladder is freed from its bed. Sometimes, we performed fundus first approach that helped us greatly to expose neck of gall bladder. Aspiration of the gall bladder helped us to grasp the fundus. A drain was put in gall bladder bed.

Outcome measures:

Primary outcomes

1. Mortality (90-day mortality and mortality at maximal follow-up).
2. Postoperative complications: early (hemorrhage, bile leak, wound infection) and late complications (biliary stricture)

4. Port site hernia Secondary outcomes

1. Conversion to open cholecystectomy.
2. Total hospital stay.
3. Intra-operative findings (duration of operation, intra-operative bleeding and iatrogenic injuries)
4. Return to work.

ELIGIBILITY:
Inclusion Criteria:

* Age: any age.
* Sex: Male and Non pregnant female.
* Patients with cardiopulmonary diseases.
* Patients who diagnose acute cholecystitis not improving on medical treatment for 48 hours.
* Patients with biliary colic, mucocele of gall bladder and pyocele of gall bladder.
* American Society of Anesthesiologist's (ASA) score: grade I, II, III.

Exclusion Criteria:

* ASA grade IV
* Patients refuse surgery.
* Documented neurological, renal and Liver disease.
* Previous percutaneous cholecystostomy
* Cases not tolerated CO2 insufflation from the start.
* Other associated problems as acute cholangitis, pancreatitis, gastro-intestinal cancer or bile duct diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
duration of operation | 2 hours
  in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No